CLINICAL TRIAL: NCT00250510
Title: A Prospective Study to Determine the Effects of a Reimbursement Incentive on Enrollment and Outcomes in a Community Weight Control Program.
Brief Title: Reimbursement Effects on Enrollment in Obesity Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Jane Fant/Assoc VP for Sponsored Research Administration, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03 DK67357 (completed); R03DK067357 (NIH)
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Obesity
Keywords: Obesity treatment; Insurance reimbursement; Health care utilization; Health care costs
MeSH Terms: conditions — Obesity; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Experimental): EatRight Program inquirers with BMI's of 30 kg/m2 or greater were told that they would have the possibility of being reimbursed 50% ($150) of their initial fee ($300) if certain conditions were met.
  Interventions: Behavioral: Simulated insurance reimbursement

INTERVENTIONS:
Behavioral: Simulated insurance reimbursement — Participants were told they would have the possibility of being reimbursed 50% ($150) of their initial fee ($300) if they: 1) paid the fee in advance or committed 3 monthly payments in advance, 2) attended 10 of 12 class sessions, and 3) lost at least 6% of their current body weight during the program.
  Arms: 2

SUMMARY:
The purpose of this study is to simulate what would occur if insurance reimbursement became available for obesity treatment but required that the individual meet defined performance milestones.

DETAILED DESCRIPTION:
This is a prospective study to determine whether a reimbursement incentive (the prospect of reimbursement of half of the out-of-pocket fee for participation in the UAB EatRight Weight Management Program, when it is contingent upon consistent Program participation and loss of 6% of initial body weight) is associated with (1) a higher rate of Program enrollment and (2) greater percent weight loss, greater reductions in medication dosages and costs, and fewer visits to health care providers after 12 weeks and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults with obesity (BMI at least 30 kg/m2)
* Commitment of the full EatRight Weight Management Program fee

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2004-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Proportion of inquirers who enroll in obesity treatment | 16 months

SECONDARY OUTCOMES:
Class attendance | 12 weeks
Percent weight loss | 12 weeks and 9 months
Changes in medication dosages and costs | 12 weeks and 9 months
Visits to health care providers | 12 weeks and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas C Heimburger, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Hubbert KA, Bussey BF, Allison DB, Beasley TM, Henson CS, Heimburger DC. Effects of outcome-driven insurance reimbursement on short-term weight control. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1423-9. doi: 10.1038/sj.ijo.0802403. PMID 14574356
- See also: UAB EatRight Weight Management Program — http://www.uab.edu/eatright